CLINICAL TRIAL: NCT03424044
Title: A Randomized, Three-way, Cross-over Study to Assess the Efficacy of a Dual-hormone Closed-loop System With XeriSol™ Glucagon vs Closed-loop System With Insulin Only vs a Predictive Low Glucose Suspend System
Brief Title: Three Way Crossover Closed Loop Study With Xeris Glucagon
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Xeris Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Jessica Castle, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17225
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Type1diabetes
Keywords: glucagon; closed-loop; Omnipod; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Dual Hormone Closed-loop Arm (Experimental): Subjects will undergo a 76 hour study with 9 hours inpatient and 67 hours outpatient using the closed-loop artificial pancreas controller in dual hormone mode and XeriSol glucagon to manage blood sugar that includes an exercise detection component that includes a reduction in insulin delivery and an increase in glucagon delivery upon detection.
  Interventions: Device: Artificial Pancreas Controller in Dual Hormone Mode; Drug: XeriSol glucagon
- Single Hormone Closed-loop Arm (Experimental): Subjects will undergo a 76 hour study with 9 hours inpatient and 67 hours outpatient using the closed-loop artificial pancreas controller in single hormone mode to manage blood sugar that includes an exercise detection component that includes a reduction in insulin delivery upon detection.
  Interventions: Device: Artificial Pancreas Controller in Single Hormone Mode
- Predictive Low Glucose Suspend Arm (Experimental): Subjects will undergo a 76 hour study with 9 hours inpatient and 67 hours outpatient using the closed-loop artificial pancreas controller in predictive low glucose suspend mode. The system will run through the closed-loop system but will utilize the patient's optimized basal rates, correction factors and carb ratios as they would normally run on their own insulin pump. But the mode will have the additional safety net of the pump suspending insulin when it predicts a hypoglycemic event.
  Interventions: Device: Artificial Pancreas Controller in Predictive Low Glucose Suspend Mode

INTERVENTIONS:
Device: Artificial Pancreas Controller in Dual Hormone Mode — The artificial pancreas controller contains an algorithm for managing blood glucose in people with type 1 diabetes which includes an exercise detection component. The algorithm has 3 modes: a single hormone closed-loop insulin only mode, a dual-hormone closed-loop insulin and glucagon mode and an insulin only mode with predictive low glucose suspend. The Closed-loop Artificial Pancreas Controller includes insulin and glucagon delivery algorithm implemented on a smart phone, utilizing sensor glucose values from a Dexcom G5 sensor and sending delivery commands to two Omnipod insulin pumps, one filled with insulin and one with glucagon.
  Arms: Dual Hormone Closed-loop Arm
Device: Artificial Pancreas Controller in Single Hormone Mode — The artificial pancreas controller contains an algorithm for managing blood glucose in people with type 1 diabetes which includes an exercise detection component. The new algorithm will have 3 modes: a single hormone closed-loop insulin only mode, a dual-hormone closed-loop insulin and glucagon mode and an insulin only mode with predictive low glucose suspend. The Closed-loop Artificial Pancreas Controller includes insulin delivery algorithm implemented on a smart phone, utilizing sensor glucose values from a Dexcom G5 sensor and sending delivery commands to one Omnipod pump filled with insulin.
  Arms: Single Hormone Closed-loop Arm
Device: Artificial Pancreas Controller in Predictive Low Glucose Suspend Mode — The artificial pancreas controller contains an algorithm for managing blood glucose in people with type 1 diabetes which includes an exercise detection component. The new algorithm will have 3 modes: a single hormone closed-loop insulin only mode, a dual-hormone closed-loop insulin and glucagon mode and an insulin only mode with predictive low glucose suspend. The Closed-loop Artificial Pancreas Controller includes insulin delivery algorithm implemented on a smart phone, utilizing sensor glucose values from a Dexcom G5 sensor and sending delivery commands to one Omnipod insulin pump filled with insulin.
  Arms: Predictive Low Glucose Suspend Arm
Drug: XeriSol glucagon — XeriSol glucagon is an investigational drug that is a stable, soluble liquid glucagon formulation that can be injected or administered through an insulin pump. XeriSol glucagon will be used to fill the Omnipod to deliver glucagon for the Artificial Pancreas Controller in Dual Hormone mode.
  Arms: Dual Hormone Closed-loop Arm

SUMMARY:
Closed-loop systems are an emerging technology that automate hormone delivery. They are quickly paving the way to revolutionize the treatment of type 1 diabetes. Several categories have emerged: dual-hormone (insulin and glucagon) closed-loop systems and closed-loop systems with insulin only, one variety of which is the low glucose suspend safety feature now available from Medtronic (MiniMed640G with SmartGuard). The study described within this protocol is designed to test the efficacy of a new closed-loop algorithm for managing blood glucose in people with type 1 diabetes before and after exercise. The new algorithm will have 3 modes: a single hormone insulin only mode, a dual-hormone insulin and glucagon mode and an insulin only mode with predictive low glucose suspend, all with an exercise detection algorithm. The purpose of this study is to determine whether a dual hormone AP using a stable investigational glucagon with an exercise detection algorithm outperforms both single hormone AP and a low glucose suspend algorithm.

DETAILED DESCRIPTION:
Subjects will undergo three approximately 76 hour studies. During each of these intervention visits, subjects will wear an Omnipod to deliver insulin and a Dexcom G5 CGM to measure glucose. In the dual-hormone closed-loop study, participants will wear a second Omnipod filled with XeriSol™ glucagon. The first day of intervention visit will be a 12 hour inpatient visit with the subsequent time spent as an outpatient. The subject will come back to the research center on Day 4 in the morning to remove all devices. The blood glucose control system is called the Artificial Pancreas Controller (APC). During one of the studies, glucose will be controlled using the dual hormone mode. During another study, glucose will be controlled using the single hormone mode. The single and dual hormone modes of the APC controller determine insulin only and insulin with glucagon delivery rates based on proportional and derivative error and contain an exercise detection component. During the other study, glucose will be controlled using a predictive low glucose suspend (PLGS) mode. In the PLGS mode, the APC will be programmed with the subject's basal profile(s) which will be transmitted to the Omnipod Personal Diabetes Manager (PDM) and allow for boluses to be inputted by the subjects for meals and corrections using their typical carb ratios and correction factors. However, this system will have a safety feature to suspend insulin delivery when sensor glucose is predicted to go below a threshold. Treatment order will be randomized.

Subjects will arrive at the clinic at approximately 7 or 8am for the inpatient visits. Subjects will eat breakfast and lunch at approximately 8:30am, noon and 6pm respectively. The dinner meal will be consumed while the subject is at home. Subjects will exercise on a treadmill for 45 minutes. Subjects will be discharged 9 hours after admission. The subject will then go home for the remainder of the study visit. Studies will be remotely monitored. Subjects will return to OHSU on Day 4 for removal of all devices.

During each study, the subject will wear one subcutaneous DexcomTM G5 continuous glucose monitoring (CGM) system. The CGM system will provide sensed glucose data every 5 minutes. The accuracy of the sensed data will be obtained by reference measurements of capillary blood glucose. Sensed glucose data will be wirelessly transmitted via Bluetooth Low Energy (BTLE) from the Dexcom G5 transmitter to the Nexus 5 master controller every five minutes. The controller for all 3 modes is a Google Nexus 5 phone. The smart phone will wirelessly communicate via BTLE to an Omnipod through a PDM (Insulet Corp. ) for automated insulin delivery or in the case of dual-hormone AP, one used for automated insulin delivery and one for automated glucagon delivery.

A physician or nurse practitioner will be present for study start-up, will be on campus for exercise on Day 1 and will be immediately available on call at all other times.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus for at least 1 year.
* Male or female subjects 21-50 years of age.
* Physically willing and able to perform 45 min of exercise.
* Current use of an insulin pump.
* Lives with another person age 18 or older who will be present while subject exercises at home and that can attend the training on using the system.
* Lives within 40 miles of OHSU main campus.
* HbA1c <= 10% at screening.
* Total daily insulin requirement is less than 139 units/day.
* Current use of a phone or other device so can be contacted by study staff off-campus.
* Willingness to follow all study procedures, including attending all clinic visits.
* Willingness to sign informed consent and HIPAA documents.

Exclusion Criteria:

* Female of childbearing potential who is pregnant or intending to become pregnant or breast-feeding, or is not using adequate contraceptive methods. Acceptable contraception includes birth control pill/patch/vaginal ring, Depo-Provera, Norplant, an IUD, the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
* Any cardiovascular disease, defined as a clinically significant EKG abnormality at the time of screening or any history of: stroke, heart failure, myocardial infarction, angina pectoris, or coronary arterial bypass graft or angioplasty. Diagnosis of 2nd and 3rd degree heart block or any non-physiological arrhythmia judged by the investigator to be exclusionary.
* Renal insufficiency (GFR < 60 ml/min, using the MDRD equation as report by the OHSU laboratory).
* Liver failure, cirrhosis, or any other liver disease that compromises liver function as determined by the investigator.
* Hematocrit of less than 36% for men, less than 32% for women.
* Hypertensive subjects with systolic blood pressure >= 160 mm Hg or diastolic blood pressure >= 100 mm Hg despite treatment or who have treatment-refractory hypertension (e.g. requiring four or more medications).
* History of severe hypoglycemia during the past 12 months prior to screening visit or hypoglycemia unawareness as judged by the investigator. Subjects will complete a hypoglycemia awareness questionnaire. Subjects will be excluded for four or more R responses.
* Adrenal insufficiency.
* Any active infection.
* Known or suspected abuse of alcohol, narcotics, or illicit drugs.
* Seizure disorder.
* Active foot ulceration.
* Severe peripheral arterial disease characterized by ischemic rest pain or severe claudication.
* Major surgical operation within 30 days prior to screening.
* Use of an investigational drug within 30 days prior to screening.
* Chronic usage of any immunosuppressive medication (such as cyclosporine, azathioprine, sirolimus, or tacrolimus).
* Bleeding disorder, treatment with warfarin, or platelet count below 50,000.
* Allergy to aspart insulin.
* Allergy to glucagon.
* Need for uninterrupted treatment of acetaminophen.
* Current administration of oral or parenteral corticosteroids.
* Any life threatening disease, including malignant neoplasms and medical history or malignant neoplasms within the past 5 years prior to screening (except basal and squamous cell skin cancer).
* Beta blockers or non-dihydropyridine calcium channel blockers.
* Current use of any medication intended to lower glucose other than insulin (e.g. use of liraglutide).
* Diagnosis of pheochromocytoma, insulinoma, or glucagonoma, personal or family history of multiple endocrine neoplasmia (MEN) 2A, MEN 2B, neurofibromatosis or von Hippel-Lindau disease.
* History of severe hypersensitivity to milk protein.
* Current use of any medication with strong anticholinergic properties, such as antihistamines, sleep aids, and antidiarrheal medications.
* Current use of indomethacin.
* Conditions that may results in low levels of releasable glucose in the liver and an inadequate reversal of hypoglycemia by glucagon such as prolonged fasting, starvation or chronic hypoglycemia as determined by the investigator.
* A positive response to any of the questions from the Physical Activity Readiness Questionnaire with one exception: subject will not be excluded if he/she takes a single blood pressure medication that doesn't impact heart rate and blood pressure is controlled on the medication (blood pressure is less than 140/90 mmHg).
* Any chest discomfort with physical activity, including pain or pressure, or other types of discomfort.
* Any clinically significant disease or disorder which in the opinion of the investigator may jeopardize the subject's safety or compliance with the protocol.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Castle, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Wilson LM, Jacobs PG, Ramsey KL, Resalat N, Reddy R, Branigan D, Leitschuh J, Gabo V, Guillot F, Senf B, El Youssef J, Steineck IIK, Tyler NS, Castle JR. Dual-Hormone Closed-Loop System Using a Liquid Stable Glucagon Formulation Versus Insulin-Only Closed-Loop System Compared With a Predictive Low Glucose Suspend System: An Open-Label, Outpatient, Single-Center, Crossover, Randomized Controlled Trial. Diabetes Care. 2020 Nov;43(11):2721-2729. doi: 10.2337/dc19-2267. Epub 2020 Sep 9. PMID 32907828

RESULTS

PARTICIPANT FLOW:
Groups:
- PLGS-SH-DH: The randomization order for subjects in this arm was predictive low glucose suspend (PLGS), single hormone (SH) and dual hormone (DH). Each visit was 76 hours and included inpatient and outpatient portions.
- DH-PLGS-SH: The randomization order for subjects in this arm was dual hormone (DH), predictive low glucose suspend (PLGS), and single hormone (SH). Each visit was 76 hours and included inpatient and outpatient portions.
- SH-DH-PLGS: The randomization order for subjects in this arm was single hormone (SH), dual hormone (DH) and predictive low glucose suspend (PLGS). Each visit was 76 hours and included inpatient and outpatient portions.
- SH-PLGS-DH: The randomization order for subjects in this arm was single hormone (SH), predictive low glucose suspend (PLGS) and dual hormone (DH). Each visit was 76 hours and included inpatient and outpatient portions.
- DH-SH-PLGS: The randomization order for subjects in this arm was dual hormone (DH), single hormone (SH) and predictive low glucose suspend (PLGS). Each visit was 76 hours and included inpatient and outpatient portions.
- PLGS-DH-SH: The randomization order for subjects in this arm was predictive low glucose suspend (PLGS), dual hormone (DH) and single hormone (SH). Each visit was 76 hours and included inpatient and outpatient portions.
- SH-SH-DH: The randomization order for this subject was single hormone (SH), dual hormone (DH) and predictive low glucose suspend (PLGS). The first SH visit wasn't completed due to technical issues and was repeated before continuing to the DH arm, which was not completed. Each visit was 76 hours and included inpatient and outpatient portions.
- SH-SH-PLGS-DH: The randomization order for this subject was single hormone (SH), predictive low glucose suspend (PLGS) and dual hormone (DH). Due to device issues, the first SH study was not completed. A second SH study was completed before continuing to PLGS and DH arms. Each arm was 76 hours and included inpatient and outpatient portions.
- DH-DH-PLGS-SH: The randomization order for this subject was dual hormone (DH), predictive low glucose suspend (PLGS) and single hormone (SH). Due to device issues, the first DH study was not completed. A second DH study was completed before continuing to PLGS and SH arms. Each arm was 76 hours and included inpatient and outpatient portions.
Period: Dexcom Training Visit (1 Week)
Arm/Group | PLGS-SH-DH | DH-PLGS-SH | SH-DH-PLGS | SH-PLGS-DH | DH-SH-PLGS | PLGS-DH-SH | SH-SH-DH | SH-SH-PLGS-DH | DH-DH-PLGS-SH
Started | 4 | 3 | 3 | 3 | 3 | 4 | 1 | 1 | 1
Completed | 4 | 3 | 3 | 3 | 3 | 4 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: First Rest Period (1-12 Weeks)
Arm/Group | PLGS-SH-DH | DH-PLGS-SH | SH-DH-PLGS | SH-PLGS-DH | DH-SH-PLGS | PLGS-DH-SH | SH-SH-DH | SH-SH-PLGS-DH | DH-DH-PLGS-SH
Started | 4 | 3 | 3 | 3 | 3 | 4 | 1 | 1 | 1
Completed | 4 | 3 | 2 | 3 | 3 | 4 | 1 | 1 | 1
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: First Intervention (76 Hours)
Arm/Group | PLGS-SH-DH | DH-PLGS-SH | SH-DH-PLGS | SH-PLGS-DH | DH-SH-PLGS | PLGS-DH-SH | SH-SH-DH | SH-SH-PLGS-DH | DH-DH-PLGS-SH
Started | 4 | 3 | 2 | 3 | 3 | 4 | 1 | 1 | 1
Completed | 4 | 3 | 2 | 3 | 2 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — device issues | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Period: Second Rest Period (7-45 Days)
Arm/Group | PLGS-SH-DH | DH-PLGS-SH | SH-DH-PLGS | SH-PLGS-DH | DH-SH-PLGS | PLGS-DH-SH | SH-SH-DH | SH-SH-PLGS-DH | DH-DH-PLGS-SH
Started | 4 | 3 | 2 | 3 | 2 | 4 | 1 | 1 | 1
Completed | 4 | 3 | 2 | 3 | 2 | 4 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (76 Hours)
Arm/Group | PLGS-SH-DH | DH-PLGS-SH | SH-DH-PLGS | SH-PLGS-DH | DH-SH-PLGS | PLGS-DH-SH | SH-SH-DH | SH-SH-PLGS-DH | DH-DH-PLGS-SH
Started | 4 | 3 | 2 | 3 | 2 | 4 | 1 | 1 | 1
Completed | 4 | 3 | 2 | 3 | 2 | 4 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Rest Period (7-45 Days)
Arm/Group | PLGS-SH-DH | DH-PLGS-SH | SH-DH-PLGS | SH-PLGS-DH | DH-SH-PLGS | PLGS-DH-SH | SH-SH-DH | SH-SH-PLGS-DH | DH-DH-PLGS-SH
Started | 4 | 3 | 2 | 3 | 2 | 4 | 1 | 1 | 1
Completed | 4 | 3 | 2 | 3 | 2 | 4 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (76 Hours)
Arm/Group | PLGS-SH-DH | DH-PLGS-SH | SH-DH-PLGS | SH-PLGS-DH | DH-SH-PLGS | PLGS-DH-SH | SH-SH-DH | SH-SH-PLGS-DH | DH-DH-PLGS-SH
Started | 4 | 3 | 2 | 3 | 2 | 4 | 1 | 1 | 1
Completed | 3 | 3 | 2 | 2 | 2 | 4 | 0 | 1 | 1
Not Completed | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Optional Fourth Rest Period (7-45 Days)
Arm/Group | PLGS-SH-DH | DH-PLGS-SH | SH-DH-PLGS | SH-PLGS-DH | DH-SH-PLGS | PLGS-DH-SH | SH-SH-DH | SH-SH-PLGS-DH | DH-DH-PLGS-SH
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Fourth Intervention Repeat Visit (76 hr)
Arm/Group | PLGS-SH-DH | DH-PLGS-SH | SH-DH-PLGS | SH-PLGS-DH | DH-SH-PLGS | PLGS-DH-SH | SH-SH-DH | SH-SH-PLGS-DH | DH-DH-PLGS-SH
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants were randomized to complete three 76 hour study visits using either dual hormone, single hormone or predictive low glucose suspend closed loop control. Treatment order was randomized
Arm/Group | All Study Participants
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Percent of Time With Sensed Glucose < 70 mg/dl
Description: Assess the percent of time that the Dexcom G5 or G6 reported sensor glucose values less than 70 mg/dl using Dexcom sensor across all three arms.
Time Frame: 4 hours post exercise on Day 1
Population: Using an intent to treat analysis, all partial and completed studies were used in this analysis. 23 subjects were randomized. One subject did not start any studies.
Measure: Median (Inter-Quartile Range); unit: percentage 4 hrs post exercise on Day 1
Groups:
- Dual Hormone Closed-loop Arm: Subjects will undergo a 76 hour study with 9 hours inpatient and 67 hours outpatient.
  Artificial Pancreas Controller in Dual Hormone Mode: The artificial pancreas controller contains an algorithm for managing blood glucose in people with type 1 diabetes which includes an exercise detection component.
  XeriSol glucagon: XeriSol glucagon is an investigational drug that is a stable, soluble liquid glucagon formulation that can be injected or administered through an insulin pump. XeriSol glucagon will be used to fill the Omnipod to deliver glucagon for the Artificial Pancreas Controller in Dual Hormone mode.
- Single Hormone Closed-loop Arm: Subjects will undergo a 76 hour study with 9 hours inpatient and 67 hours outpatient.
  Artificial Pancreas Controller in Single Hormone Mode: The artificial pancreas controller contains an algorithm for managing blood glucose in people with type 1 diabetes which includes an exercise detection component.
- Predictive Low Glucose Suspend Arm: Subjects will undergo a 76 hour study with 9 hours inpatient and 67 hours outpatient. The system will utilize the patient's optimized basal rates, correction factors and carb ratios as they would normally run but the mode will have the additional safety net of the pump suspending insulin when it predicts a hypoglycemic event.
  Artificial Pancreas Controller in Predictive Low Glucose Suspend Mode: The artificial pancreas controller contains an algorithm for managing blood glucose in people with type 1 diabetes which includes an exercise detection component.
Arm/Group | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Predictive Low Glucose Suspend Arm
Number analyzed (Participants) | 22 | 21 | 20
percentage 4 hrs post exercise on Day 1 | 0 [0 to 4.2] | 8.3 [0 to 12.5] | 4.2 [0 to 9.4]

2. Secondary Outcome: Percent of Time With Sensed Glucose Between 70-180 mg/dl
Description: Assess the percent of time that the Dexcom G5 or G6 reported sensor glucose values between 70-180 mg/dl using Dexcom sensor across all three arms.
Time Frame: entire 76 hour study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of 76 hours
Arm/Group | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Predictive Low Glucose Suspend Arm
Number analyzed (Participants) | 22 | 21 | 20
percentage of 76 hours | 71.0 (9.2) | 72.6 (9.2) | 63.4 (16.6)

3. Secondary Outcome: Number of Carbohydrate Treatments
Description: Assess the number of rescue carbohydrate treatments across all three arms per day.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of carbohydrate treatments/day
Arm/Group | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Predictive Low Glucose Suspend Arm
Number analyzed (Participants) | 22 | 21 | 20
number of carbohydrate treatments/day | 0.6 (0.9) | 1.7 (2.0) | 1.4 (1.3)

4. Secondary Outcome: Percent of Time With Sensed Glucose < 54 mg/dl
Description: Assess the percent of time that the Dexcom G5 or G6 reported sensor glucose values less than 54 mg/dl using Dexcom sensor across all three arms.
Time Frame: entire 76 hour study
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of 76 hours
Arm/Group | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Predictive Low Glucose Suspend Arm
Number analyzed (Participants) | 22 | 21 | 20
percentage of 76 hours | 0 [0 to 0.2] | 0.2 [0 to 0.8] | 0.1 [0 to 0.8]

5. Secondary Outcome: Percent of Time With Sensed Glucose > 180 mg/dl
Description: Assess the percent of time that the Dexcom G5 or G6 reported sensor glucose values greater than 180 mg/dl using Dexcom sensor across all three arms.
Time Frame: entire 76 hour study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of 76 hours
Arm/Group | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Predictive Low Glucose Suspend Arm
Number analyzed (Participants) | 22 | 21 | 20
percentage of 76 hours | 28.2 (9.4) | 25.1 (9.0) | 34.7 (16.7)

6. Secondary Outcome: Mean Amount of Insulin Delivered in One Day
Description: Assess the mean amount of insulin delivered in units/kg as documented through the artificial pancreas controller across all three arms.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units/kg/day
Arm/Group | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Predictive Low Glucose Suspend Arm
Number analyzed (Participants) | 22 | 21 | 20
units/kg/day | 42.3 (16.9) | 41.1 (16.4) | 44.0 (15.3)

7. Secondary Outcome: Mean Amount of Glucagon Delivered in One Day
Description: Assess the mean amount of XeriSol glucagon delivered in mcg/kg as documented through the artificial pancreas controller in dual hormone arm.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/kg/day
Groups:
- Dual Hormone Closed Loop: Subjects will undergo a 76 hour study with 9 hours inpatient and 67 hours outpatient.
  Artificial Pancreas Controller in Dual Hormone Mode: The artificial pancreas controller contains an algorithm for managing blood glucose in people with type 1 diabetes which includes an exercise detection component.
  XeriSol glucagon: XeriSol glucagon is an investigational drug that is a stable, soluble liquid glucagon formulation that can be injected or administered through an insulin pump. XeriSol glucagon will be used to fill the Omnipod to deliver glucagon for the Artificial Pancreas Controller in Dual Hormone mode.
Arm/Group | Dual Hormone Closed Loop
Number analyzed (Participants) | 22
mcg/kg/day | 4.5 (1.9)

ADVERSE EVENTS:
Time Frame: 13 months
Description: All participants that began/started the Dexcom training visit or a PLGS, SH, or DH arm are included in the adverse events. The numbers from the participant flow indicate that 23 subjects began the Dexcom training visit, 20 subjects began a PLGS visit, 21 subjects began a SH visit and 22 subjects began a DH visit.
Groups:
- Dexcom Training Period Arm: Subjects used the Dexcom G6 CGM along with the APC app. Subjects attended a training visit on using the Dexcom G6. Subjects used the G6 at home over the next 7 days.
Arm/Group | Dual Hormone Closed-loop Arm | Single Hormone Closed-loop Arm | Predictive Low Glucose Suspend Arm | Dexcom Training Period Arm
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/20 | 0/23
Other Adverse Events (participants affected / at risk) | 7/22 | 3/21 | 3/20 | 0/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dual Hormone Closed-loop Arm (N=22) | Single Hormone Closed-loop Arm (N=21) | Predictive Low Glucose Suspend Arm (N=20) | Dexcom Training Period Arm (N=23)
GI upset (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Burning at glucagon site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritation at zephyr site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Bruised tailbone (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Swelling at sensor site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT03424044/Prot_SAP_000.pdf